CLINICAL TRIAL: NCT01362049
Title: Mechanisms of Specific Trunk Exercises in Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sharon M. Henry, Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHRMS 10-045; 5R01HD040909-07 (NIH)
Record Dates: First submitted 2011-05-24; First posted 2011-05-27 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Low Back Pain
Keywords: Stabilization exercise; Physical therapy; Rehabilitation; Movement System Impairment exercise
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 'Eligible' Subject Group - STAB (Active Comparator): Subjects between the ages of 21-55 years with low back pain >12 months who are eligible for Treatment-Based Classification (TBC) stabilization exercises based on current criteria:
  1. straight leg raise > 90 degrees
  2. aberrant trunk movement with trunk forward flexion
  3. positive prone instability test AND/OR
  4. passive lumbar mobility testing that is judged to be hypermobile at any level.
  Interventions: Other: Physical Therapy rehabilitation: Stabilization exercises.
- 'Ineligible' Subject Group - STAB (Active Comparator): Subjects between the ages of 21-55 years with low back pain >12 months who are not eligible for the TBC-based stabilization exercises based on current criteria
  Interventions: Other: Physical Therapy rehabilitation: Stabilization exercises.
- 'Eligible' Subject Group - MSI (Active Comparator): Subjects between the ages of 21-55 years with low back pain >12 months who are eligible for Treatment-Based Classification (TBC) stabilization exercises based on current criteria:
  1. straight leg raise > 90 degrees
  2. aberrant trunk movement with trunk forward flexion
  3. positive prone instability test AND/OR
  4. passive lumbar mobility testing that is judged to be hypermobile at any level.
  Interventions: Other: Physical Therapy rehabilitation. Movement System Impairment (MSI) classification based exercise
- 'Ineligible' Subject Group -MSI (Active Comparator): Subjects between the ages of 21-55 years with low back pain >12 months who are not eligible for the TBC-based stabilization exercises based on current criteria
  Interventions: Other: Physical Therapy rehabilitation. Movement System Impairment (MSI) classification based exercise

INTERVENTIONS:
Other: Physical Therapy rehabilitation: Stabilization exercises. — The stabilization exercise protocol consists of exercises focused on improving the ability of trunk muscles to stabilize the spine, beginning with training to isolate the deeper abdominal muscles and then incorporation of these isolated contractions into other exercises. The exercise protocol progresses to include trunk flexion and extension strengthening exercises as well as abdominal bracing exercises in supine and quadruped positions, and finally to exercises in more functional positions.
  Other Names: Trunk stabilization exercises; Segmental stabilization exercises
  Arms: 'Eligible' Subject Group - STAB; 'Ineligible' Subject Group - STAB
Other: Physical Therapy rehabilitation. Movement System Impairment (MSI) classification based exercise — The MSI-classification based approach focuses on education and instruction for modifying movement strategies during functional activities, and on exercises that are specific to the classification category. First there is an analysis of and instruction in modifying a subject's direction-specific alignment and movement strategies during symptomatic functional activities. Second, there is education about the principles of tissue injury and healing, and how cumulative tissue stress contributes to microtrauma and LBP. Unique to the education process is the emphasis on how using one's particular movement strategies during functional activities may accelerate tissue stress accumulation because the strategies are used repetitively. Thirdly, there is exercise prescription that includes practice in performing modified versions of the direction-specific impairment tests from the physical exam, with an emphasis on impairments that can be modified to eliminate LBP symptoms.
  Other Names: Specific exercise; Sarhmann exercise approach; MSI exercises
  Arms: 'Eligible' Subject Group - MSI; 'Ineligible' Subject Group -MSI

SUMMARY:
The research objective is to determine which physical therapy (PT) treatment is the most efficacious for patients with lower back pain (LBP), who have been subgrouped based on certain clinical features. There is only limited evidence that supports any one PT treatment for patients with LBP since PT treatment outcomes for exercise protocols are equivocal, given the heterogeneous clinical features of patients with LBP. Thus, classification of patients with LBP into subgroups with shared clinical features has been identified as a research priority by several groups in order to prescribe the most efficacious PT treatment for each homogeneous subgroup. The investigators hypothesize that particular PT treatments are most efficacious when applied to patients with LBP, who present with particular clinical and neuromuscular features.

DETAILED DESCRIPTION:
The proposed studies focus on 2 schemas to classify LBP: 1) the Treatment-Based Classification (TBC) system, from which clinical prediction rules about who is most likely to benefit from spinal stabilization exercises (among others) have been developed, and 2) the Movement System Impairment-Based Classification (MSI) system, which includes 5 classifications of LBP named for the specific direction(s) of movements and alignments associated with the person's LBP.

The primary purpose of this proposal is to conduct a prospective, randomized, controlled Phase II clinical trial in order to examine whether or not treatment matched to a patient's specific signs and symptoms (patient-matched) per the TBC is more effective than the MSI system for improving short- (6 weeks) and long-term (12 and 24 months) outcomes in people with chronic LBP. A secondary purpose is to identify prognostic factors that predict clinical outcomes in the 2 treatment groups being compared.

Subjects will be assigned to one of two study arms:

1. eligible for Treatment-Based Classification (TBC) stabilization exercises based on current criteria ('Eligible' Subject Group); and
2. subjects who are not eligible for the TBC-based stabilization exercises ('Ineligible' Subject Group).

Within in each study arm, subjects will be randomly assigned to 1 of 2 exercise protocols for a 6-week period:

1. stabilization - a protocol focused on improving the motor control of trunk muscles to stabilize the spine; or
2. MSI-based - a classification-specific treatment focused on education and instruction for modifying movement strategies during functional activities, and on exercises specific to the classification category.

Laboratory measures (muscle activation, kinematics, forces) during standardized tasks will quantify neuromuscular impairments associated with LBP and clinical questionnaires will quantify changes in pain, function, and health status pre- and post-treatment. The addition of neuromuscular measures to these classification schemas could improve the sensitivity and specificity of each.

ELIGIBILITY:
Inclusion Criteria:

* a history of chronic LBP with or without recurrences for a minimum of 12 months;
* between 21 - 55 years of age;
* able to stand and walk without assistance;
* have an Oswestry Disability Score of 19% or higher AND/OR less than an 8 on one activity reported on the Patient Specific Functional Scale,

Exclusion Criteria:

* any major structural spinal deformity including scoliosis, kyphosis, or stenosis;
* spinal fracture or dislocation;
* osteoporosis;
* ankylosing spondylitis;
* rheumatoid arthritis;
* disc herniation with corroborating clinical signs and symptoms;
* serious spinal complications such as tumor or infection;
* previous spinal surgery;
* frank neurological loss, i.e., weakness and sensory loss;
* pain or paresthesia below the knee;
* etiology of LBP other than the lumbar spine, e.g., hip joint;
* history of neurological disease which required hospitalization;
* active treatment for cancer;
* history of unresolved cancer;
* pregnancy or less than 6 months post-partum or less than 6 months post weaning;
* magnified symptom-behavior;
* worker's compensation or disability case;
* in litigation for the LBP problem;
* have a BMI ≥ 30.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon M Henry, PT, PhD, Principal Investigator — University of Vermont
Locations (1):
- Human Motion Analysis Lab, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jacobs JV, Roy CL, Hitt JR, Popov RE, Henry SM. Neural mechanisms and functional correlates of altered postural responses to perturbed standing balance with chronic low back pain. Neuroscience. 2016 Dec 17;339:511-524. doi: 10.1016/j.neuroscience.2016.10.032. Epub 2016 Oct 19. PMID 27771534
- [Background] Boucher JA, Preuss R, Henry SM, Dumas JP, Lariviere C. The effects of an 8-week stabilization exercise program on lumbar movement sense in patients with low back pain. BMC Musculoskelet Disord. 2016 Jan 14;17:23. doi: 10.1186/s12891-016-0875-4. PMID 26762185
- [Background] Mehta R, Cannella M, Henry SM, Smith S, Giszter S, Silfies SP. Trunk Postural Muscle Timing Is Not Compromised In Low Back Pain Patients Clinically Diagnosed With Movement Coordination Impairments. Motor Control. 2017 Apr;21(2):133-157. doi: 10.1123/mc.2015-0049. Epub 2016 Aug 19. PMID 26623551
- [Background] Jacobs JV, Lomond KV, Hitt JR, DeSarno MJ, Bunn JY, Henry SM. Effects of low back pain and of stabilization or movement-system-impairment treatments on induced postural responses: A planned secondary analysis of a randomised controlled trial. Man Ther. 2016 Feb;21:210-9. doi: 10.1016/j.math.2015.08.006. Epub 2015 Aug 21. PMID 26324322
- [Background] Henry SM, Van Dillen LR, Trombley AR, Dee JM, Bunn JY. Reliability of novice raters in using the movement system impairment approach to classify people with low back pain. Man Ther. 2013 Feb;18(1):35-40. doi: 10.1016/j.math.2012.06.008. Epub 2012 Jul 15. PMID 22796388
- [Background] Lariviere C, Gagnon D, De Oliveira E Jr, Henry SM, Mecheri H, Dumas JP. Reliability of ultrasound measures of the transversus abdominis: effect of task and transducer position. PM R. 2013 Feb;5(2):104-13. doi: 10.1016/j.pmrj.2012.11.002. Epub 2013 Jan 10. PMID 23313039
- [Background] Lariviere C, Gagnon D, De Oliveira E Jr, Henry SM, Mecheri H, Dumas JP. Ultrasound measures of the lumbar multifidus: effect of task and transducer position on reliability. PM R. 2013 Aug;5(8):678-87. doi: 10.1016/j.pmrj.2013.03.010. Epub 2013 Mar 15. PMID 23507347
- [Background] Zielinski KA, Henry SM, Ouellette-Morton RH, DeSarno MJ. Lumbar multifidus muscle thickness does not predict patients with low back pain who improve with trunk stabilization exercises. Arch Phys Med Rehabil. 2013 Jun;94(6):1132-8. doi: 10.1016/j.apmr.2012.12.001. Epub 2012 Dec 7. PMID 23228626
- [Background] Henry SM, Fritz JM, Trombley AR, Bunn JY. Reliability of a treatment-based classification system for subgrouping people with low back pain. J Orthop Sports Phys Ther. 2012 Sep;42(9):797-805. doi: 10.2519/jospt.2012.4078. Epub 2012 Jun 7. PMID 22677525
- [Result] Lomond KV, Jacobs JV, Hitt JR, DeSarno MJ, Bunn JY, Henry SM. Effects of low back pain stabilization or movement system impairment treatments on voluntary postural adjustments: a randomized controlled trial. Spine J. 2015 Apr 1;15(4):596-606. doi: 10.1016/j.spinee.2014.10.020. Epub 2014 Oct 29. PMID 25452017
- [Result] Henry SM, Van Dillen LR, Ouellette-Morton RH, Hitt JR, Lomond KV, DeSarno MJ, Bunn JY. Outcomes are not different for patient-matched versus nonmatched treatment in subjects with chronic recurrent low back pain: a randomized clinical trial. Spine J. 2014 Dec 1;14(12):2799-810. doi: 10.1016/j.spinee.2014.03.024. Epub 2014 Mar 22. PMID 24662210
- [Result] Lomond KV, Henry SM, Jacobs JV, Hitt JR, Horak FB, Cohen RG, Schwartz D, Dumas JA, Naylor MR, Watts R, DeSarno MJ. Protocol to assess the neurophysiology associated with multi-segmental postural coordination. Physiol Meas. 2013 Oct;34(10):N97-105. doi: 10.1088/0967-3334/34/10/N97. Epub 2013 Sep 25. PMID 24065623

RESULTS

PARTICIPANT FLOW:
Groups:
- 'Eligible' Subject Group - MSI Treatment: Subjects between the ages of 21-55 years with low back pain >12 months who are eligible for Treatment-Based Classification (TBC) stabilization exercises based on current criteria:
  1. straight leg raise > 90 degrees
  2. aberrant trunk movement with trunk forward flexion
  3. positive prone instability test AND/OR
  4. passive lumbar mobility testing that is judged to be hypermobile at any level. Received MSI match treatment
- 'Eligible' Subject Group - STAB Treatment: Subjects between the ages of 21-55 years with low back pain >12 months who are eligible for Treatment-Based Classification (TBC) stabilization exercises based on current criteria:
  1. straight leg raise > 90 degrees
  2. aberrant trunk movement with trunk forward flexion
  3. positive prone instability test AND/OR
  4. passive lumbar mobility testing that is judged to be hypermobile at any level. Received STAB treatment
- 'Ineligible' Subject Group - MSI Treatment: Subjects between the ages of 21-55 years with low back pain >12 months who are not eligible for the TBC-based stabilization exercises based on current criteria.
  Received MSI- matched treatment
- 'Ineligible' Subject Group - STAB Treatment: Subjects between the ages of 21-55 years with low back pain >12 months who are not eligible for the TBC-based stabilization exercises based on current criteria.
  Received STAB treatment
Period: Follow-Up at 7 Weeks
Arm/Group | 'Eligible' Subject Group - MSI Treatment | 'Eligible' Subject Group - STAB Treatment | 'Ineligible' Subject Group - MSI Treatment | 'Ineligible' Subject Group - STAB Treatment
Started (Subjects who signed consent forms) | 26 | 19 | 32 | 25
Randomized and Started PT Treatment | 26 | 18 | 32 | 25
Completed | 23 | 16 | 30 | 24
Not Completed | 3 | 3 | 2 | 1
Not completed — Lost to Follow-up | 3 | 3 | 2 | 1
Period: Follow-Up at 52 Weeks (12 Months)
Arm/Group | 'Eligible' Subject Group - MSI Treatment | 'Eligible' Subject Group - STAB Treatment | 'Ineligible' Subject Group - MSI Treatment | 'Ineligible' Subject Group - STAB Treatment
Started | 23 | 16 | 30 | 24
Completed | 18 | 13 | 28 | 21
Not Completed | 5 | 3 | 2 | 3
Not completed — Lost to Follow-up | 5 | 3 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- 'Eligible' Subject Group - MSI Treatment: Subjects between the ages of 21-55 years with low back pain >12 months who are eligible for Treatment-Based Classification (TBC) stabilization exercises based on current criteria:
  1. straight leg raise > 90 degrees
  2. aberrant trunk movement with trunk forward flexion
  3. positive prone instability test AND/OR
  4. passive lumbar mobility testing that is judged to be hypermobile at any level. Received MSI-match treatment
- 'Ineligible' Subject Group - MSI Treatment: Subjects between the ages of 21-55 years with low back pain >12 months who are not eligible for the TBC-based stabilization exercises based on current criteria.
  Received MSI-match treatment
- Total: Total of all reporting groups
Arm/Group | 'Eligible' Subject Group - MSI Treatment | 'Eligible' Subject Group - STAB Treatment | 'Ineligible' Subject Group - MSI Treatment | 'Ineligible' Subject Group - STAB Treatment | Total
Number analyzed (Participants) | 26 | 19 | 32 | 25 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 26 | 19 | 32 | 25 | 102
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (11.4) | 37.1 (11.4) | 44.1 (9.4) | 45.9 (8.8) | 41.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 12 | 10 | 51
  Male | 9 | 7 | 20 | 15 | 51
Region of Enrollment [Number; unit: participants]
  United States | 26 | 19 | 32 | 25 | 102

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Oswestry Disability Scale (0-100%)
Description: Disability; Sacle 0-100% Lower score is considered better/improved
Time Frame: Baseline and 7 weeks
Population: Participants with available data are included
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 'Eligible' Subject Group - MSI: Subjects between the ages of 21-55 years with low back pain >12 months who are eligible for Treatment-Based Classification (TBC) stabilization exercises based on current criteria and who received MSI exercises for treatment
- 'Eligible' Subject Group - STAB: Subjects between the ages of 21-55 years with low back pain >12 months who are eligible for Treatment-Based Classification (TBC) stabilization exercises based on current criteria:
  1. straight leg raise > 90 degrees
  2. aberrant trunk movement with trunk forward flexion
  3. positive prone instability test AND/OR
  4. passive lumbar mobility testing that is judged to be hypermobile at any level.
  Physical Therapy rehabilitation: Stabilization exercises.: The stabilization exercise protocol consists of exercises focused on improving the ability of trunk muscles to stabilize the spine, beginning with training to isolate the deeper abdominal muscles and then incorporation of these isolated contractions into other exercises. The exercise protocol progresses to include trunk flexion and extension strengthening exercises as well as abdominal bracing exercises in supine and quadruped positions, and finally to exercises in more functional positions.
- 'Ineligible' Subject Group -MSI: Subjects between the ages of 21-55 years with low back pain >12 months who are not eligible for the TBC-based stabilization exercises based on current criteria and who received MSI exercises for treatment.
Arm/Group | 'Eligible' Subject Group - MSI | 'Eligible' Subject Group - STAB | 'Ineligible' Subject Group -MSI | 'Ineligible' Subject Group - STAB
Number analyzed (Participants) | 23 | 16 | 30 | 23
units on a scale | -8.26 (7.94) | -7.75 (8.54) | -8.00 (10.47) | -9.48 (12.02)

2. Primary Outcome: Change From Baseline in Oswestry Disability Scale (0-100%)
Description: Disability; Sacle 0-100% Lower score is considered better/improved
Time Frame: Baseline and 12 Months
Population: Participants with available data are included
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 'Eligible' Subject Group - MSI: Subjects between the ages of 21-55 years with low back pain >12 months who are eligible for Treatment-Based Classification (TBC) stabilization exercises based on current criteria and who received MSI exercises.
- 'Ineligible' Subject Group -MSI: Subjects between the ages of 21-55 years with low back pain >12 months who are not eligible for the TBC-based stabilization exercises based on current criteria and who received MSI exercises.
Arm/Group | 'Eligible' Subject Group - MSI | 'Eligible' Subject Group - STAB | 'Ineligible' Subject Group -MSI | 'Ineligible' Subject Group - STAB
Number analyzed (Participants) | 18 | 13 | 28 | 20
units on a scale | -8.8 (13.8) | -14.2 (8.9) | -10.1 (9.9) | -9.7 (11.2)

3. Primary Outcome: Change From Baseline in Numeric Pain Rating Scale (0-10 Points)
Description: Current Pain Scale 0-10 Lower score is better/improved
Time Frame: Baseline and 7 weeks
Population: Participants with available data are included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 'Eligible' Subject Group - MSI | 'Eligible' Subject Group - STAB | 'Ineligible' Subject Group -MSI | 'Ineligible' Subject Group - STAB
Number analyzed (Participants) | 21 | 14 | 30 | 25
units on a scale | -.62 (2.56) | -1 (1.62) | -1.50 (1.61) | -.92 (1.55)

4. Primary Outcome: Change From Baseline in Numeric Pain Rating Scale (0-10 Points)
Description: Current Pain Scale 0-10 Lower score is better/improved
Time Frame: Baseline and 12 months
Population: Participants with available data are included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 'Eligible' Subject Group - MSI | 'Eligible' Subject Group - STAB | 'Ineligible' Subject Group -MSI | 'Ineligible' Subject Group - STAB
Number analyzed (Participants) | 17 | 9 | 23 | 20
units on a scale | .18 (3.68) | -1.56 (1.94) | -1.35 (2.06) | -1.25 (1.33)

5. Secondary Outcome: Change From Baseline in SF-36 Health Survey (0 - 100 Points)
Description: Quality of Life - Physical Component Scale: 0-100 Higher score defines a more favorable health state
Time Frame: Baseline and 7 weeks
Population: Participants with available data are included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 'Eligible' Subject Group - MSI | 'Eligible' Subject Group - STAB | 'Ineligible' Subject Group -MSI | 'Ineligible' Subject Group - STAB
Number analyzed (Participants) | 21 | 15 | 30 | 24
units on a scale | 4.40 (6.27) | 3.99 (5.99) | 3.34 (4.87) | 1.32 (6.09)

6. Secondary Outcome: Change From Baseline in SF-36 Health Survey (0-100 Points)
Description: Quality of Life - Physical Component Scale: 0-100 Higher score defines a more favorable health state
Time Frame: Baseline and 12 months
Population: Participants with available data are included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 'Eligible' Subject Group - MSI | 'Eligible' Subject Group - STAB | 'Ineligible' Subject Group -MSI | 'Ineligible' Subject Group - STAB
Number analyzed (Participants) | 16 | 13 | 28 | 20
units on a scale | 3.16 (4.48) | 5.68 (6.25) | 2.72 (6.11) | 2.97 (6.78)

7. Secondary Outcome: Change From Baseline in Fear Avoidance Belief Questionnaire (Physical Activity Subscale 0-24 Points)
Description: fear-avoidance beliefs about physical activity Scale for Physical Activity 0-24; sum items 2, 3, 4, 5. Higher score indicates higher fear beliefs about physical acitivty
Time Frame: Baseline and 7 weeks
Population: Participants with available data are included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 'Eligible' Subject Group - MSI | 'Eligible' Subject Group - STAB | 'Ineligible' Subject Group -MSI | 'Ineligible' Subject Group - STAB
Number analyzed (Participants) | 23 | 16 | 30 | 25
units on a scale | -0.65 (3.8) | -0.53 (3.8) | -0.5 (5.2) | -1.15 (5.1)

8. Secondary Outcome: Change From Baseline in Fear Avoidance Belief Questionnaire (Physical Activity Subscale 0-24 Points)
Description: as for outcome 7
Time Frame: Baseline and 12 months
Population: Participants with available data are included
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | 'Eligible' Subject Group - MSI | 'Eligible' Subject Group - STAB | 'Ineligible' Subject Group -MSI | 'Ineligible' Subject Group - STAB
Number analyzed (Participants) | 18 | 12 | 28 | 20
units on a scale | -3.1 (4.8) | 0.6 (4.5) | -2.9 (5.3) | -1.6 (6.1)

ADVERSE EVENTS:
Time Frame: Baseline, 7 weeks, 1 year (12 months)
Groups:
- 'Eligible' Subject Group - MSI Treatment: Subjects between the ages of 21-55 years with low back pain >12 months who are eligible for Treatment-Based Classification (TBC) stabilization exercises based on current criteria:
  1. straight leg raise > 90 degrees
  2. aberrant trunk movement with trunk forward flexion
  3. positive prone instability test AND/OR
  4. passive lumbar mobility testing that is judged to be hypermobile at any level. Received MSI-matched treatment
- 'Eligible' Subject Group - STAB: Subjects between the ages of 21-55 years with low back pain >12 months who are eligible for Treatment-Based Classification (TBC) stabilization exercises based on current criteria:
  1. straight leg raise > 90 degrees
  2. aberrant trunk movement with trunk forward flexion
  3. positive prone instability test AND/OR
  4. passive lumbar mobility testing that is judged to be hypermobile at any level. Received STAB treatment
- 'Ineligible' Subject Group - MSI Treatment: Subjects between the ages of 21-55 years with low back pain >12 months who are not eligible for the TBC-based stabilization exercises based on current criteria Received MSI-matched treatment
Arm/Group | 'Eligible' Subject Group - MSI Treatment | 'Eligible' Subject Group - STAB | 'Ineligible' Subject Group - MSI Treatment | 'Ineligible' Subject Group - STAB Treatment
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/18 | 0/32 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/18 | 0/32 | 0/25
Other Adverse Events (participants affected / at risk) | 0/26 | 0/18 | 0/32 | 0/25

LIMITATIONS AND CAVEATS:
The sample size was relatively small, providing adequate power for only comparing the matched to unmatched treatments (and not the stabilization vs. Movement System Impairment exercises).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No